CLINICAL TRIAL: NCT03412019
Title: A Randomized Controlled Trial of Music vs. No Music During Cesarean Delivery on Patient Satisfaction
Brief Title: Music vs. No Music During Cesarean Delivery on Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12718
Record Dates: First submitted 2018-01-12; First posted 2018-01-26 (Actual); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Patient Satisfaction
Keywords: Music; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: There will be two arms of this randomized controlled trial as follows:
  * Control group: baseline hemodynamics and anxiety screen; no music
  * Intervention group - Mozart: A study investigator will turn on a playlist of pre-selected Mozart music.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): baseline hemodynamics and anxiety screen; no music. Satisfaction will be measured.
- Intervention group - Mozart (Experimental): A study investigator will turn on a playlist of pre-selected Mozart music. Hemodynamics and anxiety screen. Satisfaction will be measured.
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — Selections of Mozart piano sonatas
  Arms: Intervention group - Mozart

SUMMARY:
Several studies have demonstrated that music can improve various outcomes during labor and delivery. However, many of these studies didn't measure satisfaction rate accurately. This study aim to assess patient satisfaction in the setting of music or no music during the cesarean delivery. The study will be conducted in the labor and delivery unit and the expected number to enroll and complete the study is 22.

DETAILED DESCRIPTION:
Background:

Several studies have demonstrated that music can improve various outcomes during labor and delivery. In particular, patient satisfaction is often measured on a simple VAS scale, where 0 is no satisfaction and 10 is the highest satisfaction. However, patient satisfaction is a complex parameter to measure, and may be affected by a number of different factors. This study will be performed on the labor and delivery unit to assess patient satisfaction with a validated, reliable, 22-question survey in the setting of music or no music during the cesarean delivery.

Although "music" is an all-encompassing term that describes sound with different pitches and rhythms that comes together as a harmonious whole, not all music is the same. Using "music" for therapeutic purposes would be the equivalent of using "antibiotics" to cure an infection; it is too general of a term, and unlikely that such a general use of music would show a valid therapeutic benefit. However, a study demonstrated that specific selections of Mozart piano sonatas, which have a specific rhythm and mode, improve patient anxiety through a biochemical mechanism (changing the plasma levels of IL-6 and epinephrine). Therefore, in this study, the term "music" will specifically means the same Mozart sonatas as described in the prior study.

Objectives:

The objective of this study is to determine the effect of music on patient satisfaction and anxiety during cesarean delivery.

The hypothesis is that parturients exposed to music during cesarean delivery will have greater overall satisfaction and less anxiety.

Study Timelines:

* Participation begins at the time of consultation for cesarean delivery on the day of surgery, where the co-investigator Dr. Dahlawi will approach the participants and ask them to sign the ICF, and it ends after the post-anesthesia check on postoperative day 1. After recruitment and consent, patients will be randomized using a computer-generated randomization scheme will be used to allocate patients to one of the arms of the study.
* The two arms of the study are as follows:

  * Control group: baseline hemodynamics and anxiety screen; no music
  * Intervention group - Mozart: A study investigator will turn on a playlist of pre-selected Mozart music.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-50 years old
* Scheduled for elective cesarean delivery
* Nulliparity
* Singleton pregnancy
* Full term fetus (≥37.0 weeks gestational age)
* Healthy fetus (no known congenital diseases at the time of surgery)
* Requesting neuraxial anesthesia for the procedure
* Able to provide informed consent

Exclusion Criteria:

* Patient refusal
* Prior history of extensive abdominal surgery
* Active labor
* Contraindication to neuraxial anesthesia
* Uncorrected coagulopathy
* Infection at the skin site of epidural placement
* Increased intracranial pressure
* Untreated hemodynamic instability
* Known hypersensitivity to local anesthetics (a.k.a. amide or ester allergy)
* Patients with impaired hearing
* Patient on anti-anxiolytic medication

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Drzymalski, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be shared upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Available for 1 year within publication.
Access Criteria: Will need to write a formal request with reason for need to access the data

REFERENCES:
- [Background] Morgan PJ, Halpern S, Lo J. The development of a maternal satisfaction scale for caesarean section. Int J Obstet Anesth. 1999 Jul;8(3):165-70. doi: 10.1016/s0959-289x(99)80132-0. PMID 15321139
- [Background] Conrad C, Niess H, Jauch KW, Bruns CJ, Hartl W, Welker L. Overture for growth hormone: requiem for interleukin-6? Crit Care Med. 2007 Dec;35(12):2709-13. doi: 10.1097/01.ccm.0000291648.99043.b9. PMID 18074473
- [Derived] Drzymalski DM, Dahlawi M, Hall RR, Ranjan S, Best CL. The effect of Mozart music on patient satisfaction during caesarean delivery: a randomised controlled trial. Anaesthesiol Intensive Ther. 2023;55(2):114-119. doi: 10.5114/ait.2023.129007. PMID 37409839

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: no music
- Intervention Group: Music: selections of Mozart piano sonatas
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Parturients scheduled for cesarean delivery
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Patients decided to withdraw from the study prematurely
  years | 36.2 (4.2) | 32.1 (6.1) | 34.2 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: patients who were not anlayzed withdrew from the study
  Participants
    Female | 10 | 10 | 20
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: those who withdrew early were not analyzed
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 6 | 6 | 12
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: This outcome will be measured using Morgan's "Maternal Satisfaction Scale for Cesarean Section" (MSSCS).
  It is a 22-item questionnaire, each item have a Likert scale from 1-7 (1 =strongly disagree, 7=strongly agree), yielding a composite (total) score ranging 22-154, representing lowest to highest satisfaction. The questionnaire will be given to participants on post-operative day one during the hours of 8am-1pm.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 10 | 10
units on a scale | 120 (22.3) | 116 (16.4)

2. Secondary Outcome: Patient Anxiety
Description: Change in anxiety before and after surgery using a numeric rating scale from 0 (no anxiety at all) to 10 (greatest anxiety)
Time Frame: Perioperatively
Measure: Mean (Standard Deviation); unit: NRS scale (0-10)
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 10 | 10
NRS scale (0-10) | 2.5 (2.6) | 2.7 (2.7)

3. Secondary Outcome: Hemodynamic Parameter (Mean Arterial Pressure, MAP)
Description: This is the post-procedure mean arterial pressure of the patients.
Time Frame: post procedure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 10 | 10
mmHg | 82.2 (24.8) | 80.4 (8.4)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Adverse events would be tympanic membrane injury. Otherwise, would not differ from the data element definitions.
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT03412019/Prot_SAP_000.pdf